CLINICAL TRIAL: NCT04445961
Title: Respiratory Mechanics and Gas Exchange in Patients With COVID-19 and Hypoxemic Acute Respiratory Failure: Multicentral Observational Study
Brief Title: Respiratory Mechanics and Gas Exchange in Patients With COVID-19 and Hypoxemic Acute Respiratory Failure
Acronym: COVID-VENT
Status: Completed | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: COVID-VENT
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-06

CONDITIONS: SARS Pneumonia
Keywords: SARS Pneumonia; ARDS; COVID-19; compliance; recruitability
MeSH Terms: conditions — COVID-19; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Respiratory mechanics measurement — Measurement of peak inspiratory pressure, plateau pressure, calculation of static compliance and driving pressure
Diagnostic Test: Gas exchange measurement — Measurement of arterial oxygen and tension and arterial dioxide tension, calculation of arterial partial oxygen tension to inspiratory oxygen fraction (PaO2/FiO2) ratio and alveolar dead space

SUMMARY:
Data on respiratory mechanics and gas exchange in acute respiratory failure in COVID-19 patients is limited. Knowledge of respiratory mechanics and gas exchange in COVID-19 can lead to different selection of mechanical ventilation strategy, reduce ventilator-associated lung injury and improve outcomes. The objective of the study is to evaluate the respiratory mechanics, lung recruitability and gas exchange in COVID-19 -associated acute respiratory failure during the whole course of mechanical ventilation - invasive or non-invasive.

DETAILED DESCRIPTION:
In December 2019, an outbreak of a novel coronavirus (SARS-CoV-2) emerged in Wuhan, China and rapidly spread worldwide. The World Health Organization (WHO) declared the outbreak a pandemic on March 11th, 2020. The clinical disease (COVID-19) results in critical illness in about 5% of patients with predominant acute respiratory failure.

The goal of the study is the evaluation of the respiratory mechanics (peak inspiratory pressure (PIP), plateau pressure (Pplat), static compliance (Cstat), driving pressure (DP) at different positive end-expiratory pressure (PEEP) levels and different tidal volumes (Vt) (6-8 ml/kg ideal body weight), lung recruitability (by change of DP and oxygenation) and gas exchange (PaO2/FiO2 ratio and alveolar dead space) in COVID-19 -associated acute respiratory failure during the whole course of mechanical ventilation - invasive or non-invasive for selection of safe and effective PEEP level, Vt, respiratory rate (RR) and inspiratory oxygen fraction (FiO2) during the whole course of mechanical ventilation - invasive or non-invasive.

This study is multicentral observational trial in 3 University clinics.

ELIGIBILITY:
Inclusion Criteria:

* all patients with COVID-19 and acute respiratory failure on invasive and noninvasive ventilation

Exclusion Criteria:

* Patients who reached the following goals at conventional oxygen therapy (oxygen flow < 15 l/min): peripheral capillary oxygen saturation(SpO2) > 93%, no visible work of auxiliary respiratory muscles, no fatigue, stable hemodynamics (no need in any catecholamines and/or life-threatening heart rhythm abnormalities),
* less than 24 ours in intensive care unit (ICU) by any reason,
* lung emphysema,
* primary lung diseases (chronic obstructive lung disease-COPD, interstitial lung diseases, etc) or tumour metastases in lungs,
* chronic decompensated diseases with extrapulmonary organ dysfunction (tumour progression, liver cirrhosis, congestive heart failure),
* atonic coma.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with COVID-19 requiring respiratory support
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2020-08-14 (Actual)

PRIMARY OUTCOMES:
Optimum positive end-expiratory pressure (PEEP) level | On day 1 during mechanical ventilation
  Positive end-expiratory pressure (PEEP) selection at minimum level with maximum static compliance and the highest peripheral capillary oxygen saturation over fraction of inspired oxygen (SpO2/FiO2)
Optimum positive end-expiratory pressure (PEEP) level | On day 7 during mechanical ventilation
  Positive end-expiratory pressure (PEEP) selection at minimum level with maximum static compliance and the highest peripheral capillary oxygen saturation over fraction of inspired oxygen (SpO2/FiO2)
Number of patients with recruitable lung | On day 1 during mechanical ventilation
  Peripheral capillary oxygen saturation (SpO2) change from 90% after recruitment maneuver (doubled tidal volume for 15 respiratory cycles) - if peripheral capillary oxygen saturation (SpO2) after recruitment maneuver more than 95%-recruitable
Number of patients with recruitable lung | On day 7 during mechanical ventilation
  Peripheral capillary oxygen saturation (SpO2) change from 90% after recruitment maneuver (doubled tidal volume for 15 respiratory cycles) - if peripheral capillary oxygen saturation (SpO2) after recruitment maneuver more than 95%-recruitable

SECONDARY OUTCOMES:
Change in alveolar dead space | On day 1, 3, 5, 7, 10, 14, 21 during mechanical ventilation
  Calculation of the alveolar dead space using end-tidal carbon dioxide measurement and arterial carbon dioxide tension measurement
Change in plethysmogram variability during recruitment maneuver | On day 1, 3, 5, 7, 10, 14, 21 during mechanical ventilation
  Measurement of plethysmogram variability before and during recruitment maneuver
Change in arterial partial oxygen tension to inspiratory oxygen fraction (PaO2/FiO2) ratio | On day 1, 3, 5, 7, 10, 14, 21 during mechanical ventilation
  Calculation of the arterial partial oxygen tension to inspiratory oxygen fraction (PaO2/FiO2) ratio using arterial oxygen tension measurement
Optimum positive end-expiratory pressure (PEEP) level | On day 3, 5, 10, 14, 21 during mechanical ventilation
  Positive end-expiratory pressure (PEEP) selection at minimum level with maximum static compliance and the highest peripheral capillary oxygen saturation over fraction of inspired oxygen (SpO2/FiO2)
Change in driving pressure with different positive end-expiratory pressure (PEEP) levels | On day 1, 3, 5, 7, 10, 14, 21 during mechanical ventilation
  Driving pressure calculation at different positive end-expiratory pressure (PEEP) levels (8, 10, 12, 14)

CONTACTS AND LOCATIONS:
Overall Officials: Andrey I Yaroshetskiy, Dr.Med.Sc., Principal Investigator — Sechenov University
Locations (3):
- Russia (3):
  - Sechenov University Clinic #1, Moscow
  - Sechenov University Clinic #3, Moscow
  - Sechenov University Clinic #4, Moscow

REFERENCES:
- [Background] Amato MB, Meade MO, Slutsky AS, Brochard L, Costa EL, Schoenfeld DA, Stewart TE, Briel M, Talmor D, Mercat A, Richard JC, Carvalho CR, Brower RG. Driving pressure and survival in the acute respiratory distress syndrome. N Engl J Med. 2015 Feb 19;372(8):747-55. doi: 10.1056/NEJMsa1410639. PMID 25693014
- [Result] Gattinoni L, Chiumello D, Caironi P, Busana M, Romitti F, Brazzi L, Camporota L. COVID-19 pneumonia: different respiratory treatments for different phenotypes? Intensive Care Med. 2020 Jun;46(6):1099-1102. doi: 10.1007/s00134-020-06033-2. Epub 2020 Apr 14. No abstract available. PMID 32291463
- [Result] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Result] Toufen Junior C, De Santis Santiago RR, Hirota AS, Carvalho ARS, Gomes S, Amato MBP, Carvalho CRR. Driving pressure and long-term outcomes in moderate/severe acute respiratory distress syndrome. Ann Intensive Care. 2018 Dec 7;8(1):119. doi: 10.1186/s13613-018-0469-4. PMID 30535520
- [Derived] Yaroshetskiy AI, Avdeev SN, Politov ME, Nogtev PV, Beresneva VG, Sorokin YD, Konanykhin VD, Krasnoshchekova AP, Merzhoeva ZM, Tsareva NA, Trushenko NV, Mandel IA, Yavorovskiy AG. Potential for the lung recruitment and the risk of lung overdistension during 21 days of mechanical ventilation in patients with COVID-19 after noninvasive ventilation failure: the COVID-VENT observational trial. BMC Anesthesiol. 2022 Mar 4;22(1):59. doi: 10.1186/s12871-022-01600-0. PMID 35246024